CLINICAL TRIAL: NCT03356886
Title: Additional Effect of Pain Neuroscience Education to Spinal Manipulative Therapy on Pain And Disability in Chronic Low Back Pain: A Randomized Clinical Trial
Brief Title: Additional Effect of Pain Neuroscience Education to Spinal Manipulative Therapy in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Thais Cristina Chaves, Professor of the Department of Neurosciences and Behavioural Sciences of the Faculty of Medicine of Ribeirão Preto, University de São Paulo - FMRP/USP, Coordinator of the Laboratory of Research in Movement and Pain (LabMovPain), University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20112017
Record Dates: First submitted 2017-11-20; First posted 2017-11-29 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain
Keywords: Chronic Low Back Pain; Pain Neuroscience Education; Spinal Manipulative Techniques; Psychosocial Factors
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The recruited subjects will be randomized through the use of randomizer software in two groups of 52 individuals: SMT group which will receive PNE + SMT interventions or SMT alone. Both groups will be assessed at baseline (before the initial treatment session) by a blinded investigator. Immediately after the end of the last session and after the one-month follow-up, the primary outcomes and secondary outcomes will be re assessed. A single blinded investigator for the interventions administered will accomplish the assessment protocol. Another trained researcher (physiotherapist trained in SMT - 8 years of clinical experience) will administer the SMT maneuvers and a third researcher will be involved in the administration of the PNE. The treatment will last at least 8 sessions. The treatment will last at least 8 sessions lasting between 20 and 30 minutes each.
Who Masked: Investigator
Masking Description: Once the patient has accepted the invitation to participate, the same researcher (FAGT) will gather the clinical assessment and determine eligibility. After this initial assessment, participants will be randomly assigned following simple computerized randomisation procedures to one of the two treatment groups through the use of cards previously placed in opaque sealed envelopes. The allocation sequence will be generated by a researcher (TCC) not involved in the assessment and interventions, and another research assistant will assign participants to interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Manipulative Technique (SMT) (Experimental): This protocol of combined manipulation and mobilization techniques was adopted in view of the previous findings of a systematic review in which the combination of thrust mobilization and non-thrust techniques showed greater (moderate) evidence for chronic low back pain when compared to each technique alone (limited evidence). In addition, the thrust manipulation will be administered at the thoracic spine considering that a previous study found no differences in pain intensity after lumbar spine high-velocity manipulation versus non-region-specific manipulation in patients with chronic low back pain.
  Interventions: Procedure: Spinal Manipulative Technique
- SMT + Pain Neuroscience Education (Active Comparator): Content: 1) Contextualization on the importance of the program; 2) Initial concepts on neuroscience and pain, 3) How context can influence pain perception; 5) human beings as a multisensory complex; 6) Pain and memory; 7) Nociception and nociceptors; 8) The incorrect concepts on pain; 9) Concepts on pain neurophysiology; 10) Types of sensitization; 11) Descending inhibitory system; 12) The danger message and the brain processing; 13) The sensitized brain and its relationship to chronic pain; 14) The contribution of other systems to pain experience; 15) How bone, muscles and nerves send sensory information all the time; 16) Fear avoidance model revisited; 17) Encouragement to change; 18) How to develop positive attitudes and 19) Concepts of gradual exposition and gradual activity
  Interventions: Procedure: Spinal Manipulative Technique; Behavioral: Pain Neuroscience Education

INTERVENTIONS:
Procedure: Spinal Manipulative Technique — 1) The application of a global low-amplitude and high-speed manipulation at the upper thoracic region between T1 and T5 levels in the dorsal decubitus position and 2) Techniques of post-anterior central mobilization applied for 30 seconds with an average of 30 repetitions in each lumbar vertebra, from L5 to L1, using grade II joint mobilization (patients positioned in the ventral decubitus position).
Behavioral: Pain Neuroscience Education — All participants in the PNE + SMT group will initially receive a workshop on PNE in which different concepts of pain neuroscience and pain reconceptualization will be discussed and a power-point presentation with metaphors and animated videos on the topic will be employed. The PNE program will be held in 2 sessions of 40 minutes each. The topics of the intervention program will be divided into four thematic topics according to Explain Pain concepts.
  Arms: SMT + Pain Neuroscience Education

SUMMARY:
Objectives: The primary objective will be to investigate the additional effect (immediate and after one-month follow up) of pain neuroscience education (PNE) to Spinal Manipulative Therapy (SMT) on primary outcomes of pain intensity and disability in patients with chronic nonspecific low back pain (CLBP).

DETAILED DESCRIPTION:
Design: This study will be a blinded randomized controlled clinical trial. Participants: One hundred and four participants with CLBP (18 and 55 years) both genders. Interventions: Individuals included will be randomized into two possible treatment arms: PNE+SMT or SMT alone. Each treatment will last for 8 sessions. The group submitted to PNE+SMT will received in the first two initial sessions an individual face-to-face PNE program of 40 minutes.Main outcome measures: Pain intensity and low back pain-related disability will be adopted as primary outcomes and as secondary outcomes we will assess fear-avoidance, pain self-efficacy and global perceived effect of improvement. The outcomes will be assessed on three occasions: pre-intervention, immediately after 8 sessions of intervention and after one-month follow-up period. All statistical analysis will be conducted following the principles of intention to treat, and the effects of treatment will be calculated using linear mixed models. Discussion: This study will help to better understand if PNE -a psychosocial cognitive intervention- will add significant effect (immediate and at follow-up) to a movement therapy protocol based on manual therapy.

ELIGIBILITY:
Inclusion Criteria:

1. who present chronic, non-specific, continuous and recurrent low back pain lasting at least three months and
2. contemplate at least three of the following criteria: 1-hip internal rotation with> 35 °; 2-lumbar spine hypomobility; 3-absence of distal knee symptoms and 4-point FABQ Work score 19.

Exclusion Criteria:

1. pregnant women;
2. red flags (neoplasia, vertebral column fracture, vertebral osteomyelitis, infection or equine tail syndrome, rheumatic diseases, diseases that compromise cognition);
3. disc herniation;
4. women in the luteal phase will be rescheduled;
5. patients with cognitive deficits evaluated according to the Mini Mental State Examination with score less than or equal to 24 points or 22 points (low education level) and
6. previous physical therapy for low back in the past year or submitted to any health/pain education strategy. Patients will be instructed to not use pain relief medications during the intervention period of this trial and if any medication be used, participants will be encouraged to report.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity after the end and at 1 month follow-up | Baseline (before the initial treatment session), Immediately after the end of the last session and after the one-month follow-up.
  The Numerical Pain Rating Scale (NPRS) used to assess pain intensity in this trial will consist in a sequence of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable".
Change in low back pain Disability after the end and at 1 month follow-up | Baseline (before the initial treatment session), Immediately after the end of the last session and after the one-month follow-up.
  The Brazilian Portuguese version of Oswestry Disability Index (ODI) will be used to assess low back pain related disability. This instrument consists of 10 items, each of which has six response options. The total score will be calculated by summing up all the points, with the largest possible sum being 50. This sum will be transformed into a percentage by multiplying it by two.

SECONDARY OUTCOMES:
Global Perceived Effect of treatment | Immediately after the end of the last session and after the one-month follow-up.
  The global perceived effect (GPE) used for this trial is an 11-point scale that ranges from -5 ("vastly worse") through 0 ("no change") to +5 ("completely recovered") and participants are asked: "Compared to when this episode first started, how would you describe your back these days?". A higher score indicates higher perception of recovery from the condition.
Change in Fear Avoidance Beliefs after the end and at 1 month follow-up | Baseline (before the initial treatment session), Immediately after the end of the last session and after the one-month follow-up.
  The fear avoidance beliefs questionnaire (FABQ) adapted for Brazilian Portuguese consists of 16 self-response items, rated on a seven-point ordinal scale from 0 (completely disagree) to 6 (completely agree). The score is obtained for each separate subscale: one that addressed the fears and beliefs of individuals in relation to work and one that addressed their fears and beliefs about physical activities. As the content of PNE included topics about fear-avoidance, the construct will be assessed. A recent systematic review showed an association between baseline fear avoidance belief and worst levels of pain and disability as treatment outcome in chronic low back pain and showed that interventions that addressed FABs were more effective than others based on biomedical concepts.

OTHER OUTCOMES:
Cognitive Performance | Baseline
  The MMSE is a tool that can be used to systematically and thoroughly assess mental status. We used the Brazilian-Portuguese version of the tool. It is an 11-question measure that tests 5 areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score is 30. A score of ≤22 is indicative of cognitive impairment. The Mini-Mental State Examination (MMSE) was used to exclude cognitive impairment.
Pain catastrophizing | Baseline
  The Pain Catastrophizing Scale (PCS) translated and validated to Brazilian Portuguese will be used. The scale is composed of 13 items staggered on 6-point ordinal scale (0-5). The total score is the sum of the items divided by the number of items answered, with the minimum score being 0 and the maximum being 5 for each item. Higher scores indicated a greater presence of catastrophic thoughts. The total score of the scale could vary between 0 and 52 points. A recent systematic review found that catastrophizing to be associated with pain and disability at follow-up in CLBP patients.
Pain Self-Efficacy Scale - PSES | Baseline
  Study participants will be evaluated on self-efficacy related to chronic pain, which can be defined as an individual's confidence he/she can successfully produce desirable results related to living with chronic pain. The Pain Self-Efficacy Scale (PSES) has 10 items which are rated on a 7-point ordinal scale (ranging from 0: "not at all confident" to 6: "completely confident"). It was adapted and validated to Brazilian Portuguese. Previous research showed an effect on self-efficacy using a PNE intervention based on metaphors compared to an intervention using cognitive-behavioral concepts.
Hospital Anxiety and Depression Scale - HADS | Baseline
  The HADS will be employed to identify anxiety disorders and depression. It was translated and validated into Portuguese. The HADS is divided into the anxiety subscale (HADS-A) and the depression subscale (HADS-D), both containing seven interspersed items. It is composed of seven items for depression and seven items for anxiety, each item including four response options ranging from 0 to 3. A cutoff of ≥8 was described with good sensitivity and specificity values (0.70-0.90) for anxiety and depression symptoms.
STarT Back Screening Tool (SBST) | Baseline
  The SBST questionnaire was translated to Brazilian Portuguese and its psychometric measurements were checked. The questionnaire is comprised of 9 items. For the purposes of scoring and classification, respondents were given answer options of "I agree" and "I disagree" for the first 8 items, which were scored 1 and 0 points, respectively. For total scores greater than 3, classification was based on the psychosocial subscale score (items 5 to 9) as follows: scores ≤3 corresponded to medium risk and scores >3 corresponded to high risk.

CONTACTS AND LOCATIONS:
Overall Officials: Thais C Chaves, Doctor, Study Chair — University São Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Geneen LJ, Martin DJ, Adams N, Clarke C, Dunbar M, Jones D, McNamee P, Schofield P, Smith BH. Effects of education to facilitate knowledge about chronic pain for adults: a systematic review with meta-analysis. Syst Rev. 2015 Oct 1;4:132. doi: 10.1186/s13643-015-0120-5. PMID 26428467
- [Background] Louw A, Puentedura EL, Mintken P. Use of an abbreviated neuroscience education approach in the treatment of chronic low back pain: a case report. Physiother Theory Pract. 2012 Jan;28(1):50-62. doi: 10.3109/09593985.2011.562602. Epub 2011 Jul 3. PMID 21721995
- [Background] Gallagher L, McAuley J, Moseley GL. A randomized-controlled trial of using a book of metaphors to reconceptualize pain and decrease catastrophizing in people with chronic pain. Clin J Pain. 2013 Jan;29(1):20-5. doi: 10.1097/AJP.0b013e3182465cf7. PMID 22688603
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Dougherty PE, Karuza J, Savino D, Katz P. Evaluation of a modified clinical prediction rule for use with spinal manipulative therapy in patients with chronic low back pain: a randomized clinical trial. Chiropr Man Therap. 2014 Nov 18;22(1):41. doi: 10.1186/s12998-014-0041-8. eCollection 2014. PMID 25426289
- [Background] Hidalgo B, Detrembleur C, Hall T, Mahaudens P, Nielens H. The efficacy of manual therapy and exercise for different stages of non-specific low back pain: an update of systematic reviews. J Man Manip Ther. 2014 May;22(2):59-74. doi: 10.1179/2042618613Y.0000000041. PMID 24976749
- [Background] Clarke CL, Ryan CG, Martin DJ. Pain neurophysiology education for the management of individuals with chronic low back pain: systematic review and meta-analysis. Man Ther. 2011 Dec;16(6):544-9. doi: 10.1016/j.math.2011.05.003. Epub 2011 Jun 25. PMID 21705261